CLINICAL TRIAL: NCT05534438
Title: Stereotactic Body Radiation Therapy (SBRT) to Extend the Benefit of Systemic Therapy in Patients With Solitary Disease Progression
Brief Title: A Study on Adding Precisely Targeted Radiation Therapy (Stereotactic Body Radiation Therapy) to the Usual Treatment Approach (Drug Therapy) in People With Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-259
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Oligometastatic Breast Carcinoma; Breast Cancer; Metastatic Breast Cancer; Metastatic Breast Carcinoma; ER+ Breast Cancer; HER2+ Breast Cancer
Keywords: oligometastatic breast cancer; breast cancer; ER+ Breast Cancer; HER2+ Breast Cancer; Metastatic Breast Cancer; Stereotactic Body Radiation Therapy; 22-259; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with oligometastatic breast cancer (Experimental): Participants with oligometastatic breast cancer with isolated progression after sustained (>=6 month) response to systemic therapy. Participants will receive image guided, SBRT to the progressive lesion identified on imaging. Participants will be maintained on their existing line of systemic therapy. Systemic therapy will be held during days of radiation and resume following completion of radiation.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — SBRT will be initiated as soon as possible, at not beyond 8 weeks of baseline measurements. Recommended dosing is per department standards for oligometastatic disease (ie, 10 Gy x 3 or 7-8 Gy x 5 fractions daily, excluding weekends and departmental holidays)
  Other Names: SBRT

SUMMARY:
The purpose of this study is to see if using Stereotactic Body Radiation Therapy/SBRT to treat a single metastatic site where cancer has worsened may be an effective treatment for people with oligometastatic breast cancer. Participants will stay on their usual drug therapy while they receive SBRT. This combination of SBRT to a single metastatic site and usual drug therapy may prevent participants' cancer from worsening in other metastatic sites or spreading.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing and able to provide informed consent
* Metastatic breast cancer, biopsy proven

  * ER+/HER2-, defined as >5% ER+ staining
  * HER2+ (regardless of ER status), including HER2-low and high expressors
* History of at least 6 months, sustained response to systemic therapy (clinically or radiographically defined as complete or stable response without progression)
* Isolated site of disease progression on FDG PET scan
* Consented to 12-245
* ECOG performance status 0-1

Exclusion Criteria:

* Pregnancy
* Serious medical comorbidity precluding radiation, including connective tissue disorders
* Intracranial disease (including previous intracranial involvement)
* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 months from start of SBRT delivery
  The primary objective is to assess progression free survival, defined as systemic progression or death, within 3 months from start of Stereotactic Body Radiation Therapy/SBRT delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Xu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org